CLINICAL TRIAL: NCT04910243
Title: The Practice of Providing Palliative Care in the Situation of the COVID-19 (Coronavirus Disease 2019) Pandemic in the Perspective of Physicians and Nurses - Survey Study
Brief Title: The Practice of Providing Palliative Care in the Situation of the COVID-19 (Coronavirus Disease 2019) Pandemic in Czech Republic
Acronym: PEOpLe-C19
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Jan Malaska, Senior Investigator, Brno University Hospital
Other Study IDs: PEOpLe-C19 study
Record Dates: First submitted 2021-05-28; First posted 2021-06-02 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Distress, Emotional
Keywords: Palliative Care; Compassionate Care; End-of-life decisions; Moral distress
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physicians: Physicians managing patients with COVID-19 admitted at ICU during period of COVID-19 pandemic.
  Interventions: Other: Questionnaire Survey
- Nurses: Nurses providing care to patients with COVID-19 admitted at ICU during period of COVID-19 pandemic.
  Interventions: Other: Questionnaire Survey

INTERVENTIONS:
Other: Questionnaire Survey — Physicians providing care to patients with COVID-19 admitted at ICU in period of COVID-19 pandemic will be questioned by electronic web-based survey within Masaryk University information system.

SUMMARY:
Pandemic of coronavirus SARS-CoV-2 (Severe Acute Respiratory Syndrome coronavirus 2) causing the disease COVID-19 (Coronavirus Disease 2019) overwhelmed healthcare and brought new challenges and stressful situations.

DETAILED DESCRIPTION:
In a short time, the capacities of intensive care units (ICU) were filled in many countries and regions. Due to the need for an excessive number of patients requiring intensive care, physicians and nurses who do not routinely provide care to critically ill patients or do not have the appropriate training (non-ICU clinician) were involved in the care of COVID-19 (Coronavirus Disease 2019) patients. In this context, ICU directly dedicated to the care of patients with COVID-19 ARDS (Acute Respiratory Distress Syndrome) were also opened. Non-ICU clinicians were more or less involved together with the standard ICU staff in palliative care, including End-of-Life decision (EOLD) making, even in a situation of limited scarce resources (equipment or personnel). New workplace and scope of work, which did not correspond to the standard activity or education, most likely led to an increased stress load. EOLD can also be one of the factors leading to increased stress levels. The aim of the project is to describe the practice of palliative care for patients with COVID-19 in a situation of pandemic COVID-19 and to identify factors leading to possible moral distress related with EOLD.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers (physicians and nurses) providing care to patients with COVID-19 admitted at ICU in period of COVID-19 pandemic.

Exclusion Criteria:

* Healthcare professionals who did not managed COVID-19 patients admitted at the ICU in situation of COVID-19 pandemic in the period 2020/2021.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare providers (physicians and nurses) providing care to patients with COVID-19 admitted at ICU in period of COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Change of practice of providing palliative care at ICU in COVID-19 pandemic | Through study completion, an average of 1 month
  Change of practice of providing palliative care including EOLD practice in patients with COVID-19 admitted at ICU during pandemic.

SECONDARY OUTCOMES:
Risk factors for moral distress | Through study completion, an average of 1 month
  Identify factors leading to moral distress during COVID-19 pandemic and describe possible different risk factors by profession

CONTACTS AND LOCATIONS:
Overall Officials: Tereza Prokopová, M.D., Principal Investigator — Masaryk University Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prokopova T, Hudec J, Vrbica K, Stasek J, Pokorna A, Stourac P, Rusinova K, Kerpnerova P, Stepanova R, Svobodnik A, Malaska J; RIPE-ICU study group. Palliative care practice and moral distress during COVID-19 pandemic (PEOpLE-C19 study): a national, cross-sectional study in intensive care units in the Czech Republic. Crit Care. 2022 Jul 19;26(1):221. doi: 10.1186/s13054-022-04066-1. PMID 35854318